CLINICAL TRIAL: NCT00005359
Title: Genetics of Asthma and Bronchial Hyperresponsiveness
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4246; R01HL048341-14 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-07

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To investigate the genetics of asthma by reexamining a carefully characterized population of patients with asthma, and by studying their families.

DETAILED DESCRIPTION:
BACKGROUND:

The development of asthma requires exposure to inciting agents such as allergens and environmental pollutants, as well as the presence of host or genetic factors. Understanding the genetics of bronchial hyperresponsiveness (BHR) and allergy will delineate mechanisms that are important in the pathogenesis and therapy of asthma. While both genetic and environmental factors and their interactions are felt to be important, their precise role is not fully understood.

DESIGN NARRATIVE:

The probands are from the 'asthma' center Beatrixoord in Haren, The Netherlands which was started in 1962. In collaboration with Dr Dirkje Postma of Holland, data are available on approximately 1200 patients who were first studied in 1963-1970 using the same protocol. Family studies of the children and grandchildren of these original probands are underway. At this time, 85 complete families have been characterized and clinical data and DNA are available for analysis in Baltimore. Families are being ascertained so that the investigators can test the fit of genetic models through segregation analyses. The major aim of the study is to identify major genes for bronchial hyperresponsiveness (BHR) and asthma by linkage with highly polymorphic DNA markers. Since allergy is commonly associated with asthma, a second goal of the study is to identify major genes for atopy using similar linkage studies. Allergic factors under study include skin test reactivity to common allergens, serum total and specific IgE levels, and blood eosinophilia. Complex segregation analysis will be performed separately for asthma, BHR and allergy. The most parsimonious model from the segregation analysis will be used for linkage analysis. Initially, candidate regions of the genome will be evaluated. Then, a systematic search of the genome will be performed using highly polymorphic informative makers. When a linkage is detected, candidate genes in that specific area will be studied.

The study was renewed in FY 1999 and in FY 2004 to: further characterize asthma and closely related phenotypes; perform genetic modeling (complex segregation analysis) using one and two locus models as well as bivariate segregation analysis; complete the genome wide screen; fine map regions of interest and identify candidate genes, perform linkage disequilibrium and haplotype sharing analyses; and perform case control analysis of susceptibility and severity candidate genes for asthma.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Meyers — Wake Forest University

REFERENCES:
- [Background] Bleecker ER, Postma DS, Meyers DA. Genetic susceptibility to asthma in a changing environment. Ciba Found Symp. 1997;206:90-9; discussion 99-105, 106-10. doi: 10.1002/9780470515334.ch6. PMID 9257007
- [Background] Levitt RC, Holroyd KJ. Fine-structure mapping of genes providing susceptibility to asthma on chromosome 5q31-q33. Clin Exp Allergy. 1995 Nov;25 Suppl 2:119-23. doi: 10.1111/j.1365-2222.1995.tb00439.x. No abstract available. PMID 8590330
- [Background] Postma DS, Bleecker ER, Amelung PJ, Holroyd KJ, Xu J, Panhuysen CI, Meyers DA, Levitt RC. Genetic susceptibility to asthma--bronchial hyperresponsiveness coinherited with a major gene for atopy. N Engl J Med. 1995 Oct 5;333(14):894-900. doi: 10.1056/NEJM199510053331402. PMID 7666875
- [Background] DiSilvestre D, Kleeberger SR, Johns J, Levitt RC. Structure and DNA sequence of the mouse MnSOD gene. Mamm Genome. 1995 Apr;6(4):281-4. doi: 10.1007/BF00352417. PMID 7613035
- [Background] Monitto CL, Levitt RC, DiSilvestre D, Holroyd KJ. Localization of the A3 adenosine receptor gene (ADORA3) to human chromosome 1p. Genomics. 1995 Apr 10;26(3):637-8. doi: 10.1016/0888-7543(95)80194-q. No abstract available. PMID 7607699
- [Background] Meyers DA, Bleecker ER. Approaches to mapping genes for allergy and asthma. Am J Respir Crit Care Med. 1995 Jul;152(1):411-3. doi: 10.1164/ajrccm.152.1.7599858. No abstract available.
- [Background] Levitt RC, Ewart SL. Genetic susceptibility to atracurium-induced bronchoconstriction. Am J Respir Crit Care Med. 1995 May;151(5):1537-42. doi: 10.1164/ajrccm.151.5.7735612.
- [Background] Levitt RC, Kiser MB, Dragwa C, Jedlicka AE, Xu J, Meyers DA, Hudson JR. Fluorescence-based resource for semiautomated genomic analyses using microsatellite markers. Genomics. 1994 Nov 15;24(2):361-5. doi: 10.1006/geno.1994.1628. PMID 7698760
- [Background] Schwengel DA, Jedlicka AE, Nanthakumar EJ, Weber JL, Levitt RC. Comparison of fluorescence-based semi-automated genotyping of multiple microsatellite loci with autoradiographic techniques. Genomics. 1994 Jul 1;22(1):46-54. doi: 10.1006/geno.1994.1344. PMID 7959791
- [Background] He P, Ma Y, Zhao G, Dai H, Li H, Chang L, Zhang Z. FaRE1: a transcriptionally active Ty1-copia retrotransposon in strawberry. J Plant Res. 2010 Sep;123(5):707-14. doi: 10.1007/s10265-009-0290-0. Epub 2009 Dec 18. PMID 20020171
- [Background] Howard TD, Bleecker ER, Stine OC. Fluorescent allele-specific PCR (FAS-PCR) improves the reliability of single nucleotide polymorphism screening. Biotechniques. 1999 Mar;26(3):380-1. doi: 10.2144/99263bm01. No abstract available. PMID 10090967
- [Background] Stine OC, Xu J, Meyers DA, Bleecker ER. Approaches to fine mapping in asthma. Clin Exp Allergy. 1998 Apr;28 Suppl 1:98-100; discussion 108-10. doi: 10.1046/j.1365-2222.1998.0280s1098.x. No abstract available. PMID 9641604
- [Background] Panhuysen CI, Bleecker ER, Koeter GH, Meyers DA, Postma DS. Characterization of obstructive airway disease in family members of probands with asthma. An algorithm for the diagnosis of asthma. Am J Respir Crit Care Med. 1998 Jun;157(6 Pt 1):1734-42. doi: 10.1164/ajrccm.157.6.9606088. PMID 9620899
- [Background] Bleecker ER, Postma DS, Meyers DA. Evidence for multiple genetic susceptibility loci for asthma. Am J Respir Crit Care Med. 1997 Oct;156(4 Pt 2):S113-6. doi: 10.1164/ajrccm.156.4.12tac7. PMID 9351590
- [Background] Bleecker ER, Amelung PJ, Levitt RC, Postma DS, Meyers DA. Evidence for linkage of total serum IgE and bronchial hyperresponsiveness to chromosome 5q: a major regulatory locus important in asthma. Clin Exp Allergy. 1995 Nov;25 Suppl 2:84-8; discussion 95-6. doi: 10.1111/j.1365-2222.1995.tb00430.x. No abstract available. PMID 8590353
- [Background] Meyers DA, Xu J, Postma DS, Levitt RC, Bleecker ER. Two locus segregation and linkage analysis for total serum IgE levels. Clin Exp Allergy. 1995 Nov;25 Suppl 2:113-5. doi: 10.1111/j.1365-2222.1995.tb00437.x. No abstract available. PMID 8590328
- [Background] Wiesch DG, Meyers DA. Strategies for analyzing genotype-phenotype relationships in asthma. J Allergy Clin Immunol. 2000 Feb;105(2 Pt 2):S482-6. doi: 10.1016/s0091-6749(00)90047-2. PMID 10669528
- [Background] Howard TD, Meyers DA, Bleecker ER. Mapping susceptibility genes for asthma and allergy. J Allergy Clin Immunol. 2000 Feb;105(2 Pt 2):S477-81. doi: 10.1016/s0091-6749(00)90046-0. PMID 10669527
- [Background] Koppelman GH, Reijmerink NE, Colin Stine O, Howard TD, Whittaker PA, Meyers DA, Postma DS, Bleecker ER. Association of a promoter polymorphism of the CD14 gene and atopy. Am J Respir Crit Care Med. 2001 Mar;163(4):965-9. doi: 10.1164/ajrccm.163.4.2004164. PMID 11282774
- [Background] Xu J, Postma DS, Howard TD, Koppelman GH, Zheng SL, Stine OC, Bleecker ER, Meyers DA. Major genes regulating total serum immunoglobulin E levels in families with asthma. Am J Hum Genet. 2000 Nov;67(5):1163-73. doi: 10.1086/321190. Epub 2000 Oct 6. PMID 11023809
- [Background] Koppelman GH, Stine OC, Xu J, Howard TD, Zheng SL, Kauffman HF, Bleecker ER, Meyers DA, Postma DS. Genome-wide search for atopy susceptibility genes in Dutch families with asthma. J Allergy Clin Immunol. 2002 Mar;109(3):498-506. doi: 10.1067/mai.2002.122235. PMID 11897998
- [Background] Xu J, Bleecker ER, Jongepier H, Howard TD, Koppelman GH, Postma DS, Meyers DA. Major recessive gene(s) with considerable residual polygenic effect regulating adult height: confirmation of genomewide scan results for chromosomes 6, 9, and 12. Am J Hum Genet. 2002 Sep;71(3):646-50. doi: 10.1086/342216. Epub 2002 Jul 15. PMID 12119602
- [Background] Howard TD, Meyers DA, Bleecker ER. Mapping susceptibility genes for allergic diseases. Chest. 2003 Mar;123(3 Suppl):363S-8S. doi: 10.1378/chest.123.3_suppl.363s-a. PMID 12628976
- [Background] Koppelman GH, Jansen DF, Schouten JP, van der Heide S, Bleecker ER, Meyers DA, Postma DS. Sibling effect on atopy in children of patients with asthma. Clin Exp Allergy. 2003 Feb;33(2):170-5. doi: 10.1046/j.1365-2222.2003.01591.x. PMID 12580908
- [Background] Howard TD, Postma DS, Jongepier H, Moore WC, Koppelman GH, Zheng SL, Xu J, Bleecker ER, Meyers DA. Association of a disintegrin and metalloprotease 33 (ADAM33) gene with asthma in ethnically diverse populations. J Allergy Clin Immunol. 2003 Oct;112(4):717-22. doi: 10.1016/s0091-6749(03)01939-0. PMID 14564349
- [Background] Jongepier H, Boezen HM, Dijkstra A, Howard TD, Vonk JM, Koppelman GH, Zheng SL, Meyers DA, Bleecker ER, Postma DS. Polymorphisms of the ADAM33 gene are associated with accelerated lung function decline in asthma. Clin Exp Allergy. 2004 May;34(5):757-60. doi: 10.1111/j.1365-2222.2004.1938.x. PMID 15144468
- [Background] Meyers DA, Postma DS, Stine OC, Koppelman GH, Ampleford EJ, Jongepier H, Howard TD, Bleecker ER. Genome screen for asthma and bronchial hyperresponsiveness: interactions with passive smoke exposure. J Allergy Clin Immunol. 2005 Jun;115(6):1169-75. doi: 10.1016/j.jaci.2005.01.070. PMID 15940130
- [Background] Postma DS, Meyers DA, Jongepier H, Howard TD, Koppelman GH, Bleecker ER. Genomewide screen for pulmonary function in 200 families ascertained for asthma. Am J Respir Crit Care Med. 2005 Aug 15;172(4):446-52. doi: 10.1164/rccm.200407-864OC. Epub 2005 May 18. PMID 15901612
- [Background] Oostendorp J, Postma DS, Volders H, Jongepier H, Kauffman HF, Boezen HM, Meyers DA, Bleecker ER, Nelemans SA, Zaagsma J, Meurs H. Differential desensitization of homozygous haplotypes of the beta2-adrenergic receptor in lymphocytes. Am J Respir Crit Care Med. 2005 Aug 1;172(3):322-8. doi: 10.1164/rccm.200409-1162OC. Epub 2005 May 5. PMID 15879418
- [Background] Teeter JG, Bleecker ER. Mechanisms of asthma. Curr Opin Pulm Med. 1996 Jan;2(1):23-8. PMID 9363111